CLINICAL TRIAL: NCT04747288
Title: Using the Objective Measurement Methods to Evaluate the Association With TCM Pattern and TCM Tongue Diagnosis for Autoimmune Disease and Dry Eye Syndrome
Brief Title: Objective Measurement With TCM Pattern for AIDDES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-12-014BC
Record Dates: First submitted 2021-02-09; First posted 2021-02-10 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Sjögren's Syndrome; Systemic Lupus Erythematosus; Dry Eye Syndrome
Keywords: Sjögren's syndrome; Systemic Lupus Erythematosus; Dry Eye Syndrome
MeSH Terms: conditions — Sjogren's Syndrome; Lupus Erythematosus, Systemic; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sjögren's syndrome: Sjögren's syndrome patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 2002 American-European Consensus Criteria for SS (AECG). Exclusion Criteria: NA.
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Diseast Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: 36-Item Short Form Survey (SF-36)
- Systemic lupus erythematosus: Systemic lupus erythematosus patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 1982 and 1997 revised Systemic lupus erythematosus criteria. Exclusion Criteria: NA.
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Diseast Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: 36-Item Short Form Survey (SF-36)
- Dry eye syndrome: Dry eye syndrome patients were screened in the ophthalmology outpatient departments, rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) Schirmer's test less than 10 mm/5 min. Exclusion Criteria: NA.
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Diseast Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: 36-Item Short Form Survey (SF-36)
- non AIDDES Healthy Controls: Non AIDDES Healthy Controls were enrolled with inclusion criteria: (1) aged between 20 and 75 years; (2) without any Chronic disease. Exclusion Criteria: any Sjögren's syndrome, Systemic lupus erythematosus, or Dry eye syndrome.
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis

INTERVENTIONS:
Diagnostic Test: Traditional Chinese Medicine pattern — Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE) for comparing with the Dry eye syndrome (DES) and non AIDDES Healthy Controls subjects will take the Traditional Chinese Medicine pattern diagnosis.
Diagnostic Test: Traditional Chinese Medicine tongue diagnosis — Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE) for comparing with the Dry eye syndrome (DES) and non AIDDES Healthy Controls subjects will take the Traditional Chinese Medicine tongue diagnosis.
Diagnostic Test: Heart rate variability — Autoimmune disease (AID) as Sjögren's syndrome (SJS) and Systemic lupus erythematosus (SLE) for comparing with the Dry eye syndrome (DES) subjects will take the Heart rate variability.
  Groups: Dry eye syndrome; Sjögren's syndrome; Systemic lupus erythematosus
Diagnostic Test: Schirmer's test — Autoimmune disease (AID) as Sjögren's syndrome (SJS) and Systemic lupus erythematosus (SLE) for comparing with the Dry eye syndrome (DES) subjects will take the Schirmer's test.
  Groups: Dry eye syndrome; Sjögren's syndrome; Systemic lupus erythematosus
Diagnostic Test: Ocular Surface Diseast Index (OSDI) — Autoimmune disease (AID) as Sjögren's syndrome (SJS) and Systemic lupus erythematosus (SLE) for comparing with the Dry eye syndrome (DES) subjects will take the Ocular Surface Diseast Index (OSDI).
  Groups: Dry eye syndrome; Sjögren's syndrome; Systemic lupus erythematosus
Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) — Autoimmune disease (AID) as Sjögren's syndrome (SJS) and Systemic lupus erythematosus (SLE) for comparing with the Dry eye syndrome (DES) subjects will take the EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI).
  Groups: Dry eye syndrome; Sjögren's syndrome; Systemic lupus erythematosus
Diagnostic Test: 36-Item Short Form Survey (SF-36) — Autoimmune disease (AID) as Sjögren's syndrome (SJS) and Systemic lupus erythematosus (SLE) for comparing with the Dry eye syndrome (DES) subjects will take the 36-Item Short Form Survey (SF-36).
  Groups: Dry eye syndrome; Sjögren's syndrome; Systemic lupus erythematosus

SUMMARY:
To explore the association with TCM pattern and TCM tongue diagnosis for Autoimmune disease and Dry eye syndrome.

DETAILED DESCRIPTION:
Objective: To explore the association with TCM pattern and TCM tongue diagnosis for Autoimmune disease and Dry eye syndrome.

Method:

This study wants to include the 1000 Autoimmune disease (AID) subjects as 800 Sjögren's syndrome (SJS) and 200 Systemic lupus erythematosus (SLE) for comparing with the 500 Dry eye syndrome (DES) subjects. AID and DES subjects will be enrolled to evaluate at V1 Baseline and follow-up for 6 times evaluation with one month interval during one year. And the non-AID-non-DES healthy control subjects will be also included in our study for comparison with the dry eye syndrome and healthy control. This study want to use objective measurement and questionnaires as TCM pattern, OSDI, ESSPRI, SF-36, Schirmer's test, TCM heart rate variability, and TCM tongue diagnosis to differentiate AID, DES and healthy control.

Expected Results:

1. To evaluate the difference among TCM pattern, OSDI, ESSPRI, SF-36, Schirmer's test, TCM heart rate variability, and TCM tongue diagnosis to differentiate between AID and DES.
2. To evaluate the difference among TCM pattern and TCM tongue diagnosis among the AID groups, DES group, and healthy control.

Keyword: Autoimmune disease, Sjögren's syndrome, Systemic lupus erythematosus, Dry eye syndrome, TCM pattern, TCM tongue diagnosis.

ELIGIBILITY:
Sjögren's syndrome

* Inclusion Criteria:

  1. aged between 20 and 75 years
  2. fulfilled the 2002 American-European Consensus Criteria for SS (AECG)
* Exclusion Criteria: NA

Systemic lupus erythematosus

* Inclusion Criteria:

  1. aged between 20 and 75 years
  2. fulfilled the 1982 and 1997 ACR revised Systemic lupus erythematosus criteria
* Exclusion Criteria: NA

Dry eye syndrome

* Inclusion Criteria:

  1. aged between 20 and 75 years
  2. Schirmer's test less than 10 mm/5 min
* Exclusion Criteria: NA

non AIDDES Healthy Controls

* Inclusion Criteria:

  1. aged between 20 and 75 years
  2. without any Chronic disease
* Exclusion Criteria: any Sjögren's syndrome, Systemic lupus erythematosus, or Dry eye syndrome.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Autoimmune disease (AID) as Sjögren's syndrome (SJS), and Dry eye syndrome (DES) subjects were screened in the ophthalmology outpatient departments, rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital.
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
TCM pattern | One year
  TCM pattern is a tool for detecting the constitution among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Dry eye syndrome (DES), and healthy control.
TCM tongue diagnosis | One year
  TCM tongue diagnosis is a tool for detecting tongue expression among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Dry eye syndrome (DES), and healthy control.
Heart rate variability (HRV) | One year
  Heart rate variability (HRV) is a tool for detecting ratio between High-frequency (HF) activity and low-frequency (LF) activity among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE),and Dry eye syndrome (DES).
Schirmer's test | One year
  Schirmer's test is a tool for evaluating aqueous tear production among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), and Dry eye syndrome (DES).
OSDI(Ocular Surface Disease Index) | One year
  OSDI is a tool to rate the severity of dry eye disease among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), and Dry eye syndrome (DES).
ESSPRI(EULAR Sjögren's Syndrome Patient Reported Index) | One year
  ESSPRI is a tool for evaluating the symptoms of SJS among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), and Dry eye syndrome (DES).
SF-36(36-Item Short Form Survey ) | One year
  SF-36 is a tool for evaluating Health-Related Quality of Life among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), and Dry eye syndrome (DES).

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ching-Mao, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Ching-Mao Chang, Taipei, Taiwan